CLINICAL TRIAL: NCT02168803
Title: A Phase 1b Study to Characterize the Pharmacokinetics of Evacetrapib and Potential for Accumulation After Dosing for 12, 24, and 52 Weeks
Brief Title: A Study of Evacetrapib in Participants With Abnormal Cholesterol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15340; I1V-MC-EIBM (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-05-22; First posted 2014-06-20 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-02

CONDITIONS: Dyslipidemia
Keywords: abnormal cholesterol
MeSH Terms: conditions — Dyslipidemias | interventions — evacetrapib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Evacetrapib: Single Dose (Experimental): Single oral dose of evacetrapib on Day 1
  Interventions: Drug: Evacetrapib
- Evacetrapib: Multiple Dose 12 Weeks (Experimental): Evacetrapib administered orally once daily beginning on Day 8 for 12 consecutive weeks
  Interventions: Drug: Evacetrapib
- Evacetrapib: Multiple Dose 24 Weeks (Experimental): Evacetrapib administered orally once daily beginning on Day 8 for 24 consecutive weeks
  Interventions: Drug: Evacetrapib
- Evacetrapib: Multiple Dose 52 Weeks (Experimental): Evacetrapib administered orally once daily beginning on Day 8 for 52 consecutive weeks
  Interventions: Drug: Evacetrapib

INTERVENTIONS:
Drug: Evacetrapib — Administered orally
  Other Names: LY2484595

SUMMARY:
The main purpose of this study is to measure how much of the drug gets into the blood stream and how long it takes the body to get rid of it when given once a day for 12, 24, and 52 weeks to participants with abnormal amounts of cholesterol and/or fat in the blood stream. Information about any side effects that may occur will also be collected.

This study will also evaluate how the study drug reacts in the body when given once a day for 12, 24 and 52 weeks and how the body responds and returns to normal when the treatment is complete. The relationship between study drug and the results from the how the study drug reacts in the body may be explored, if needed.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy participants or have stable medical conditions that, in the investigator's opinion, will not significantly alter the disposition of the drug, will not place the participant at increased risk by participating in the study, and will not interfere with interpretation of the data and meets one of the following criteria:

  * Elevated low-density lipoprotein cholesterol (LDL-C) greater than 100 milligrams per deciliter (mg/dL), OR
  * Low high-density lipoprotein cholesterol (HDL-C) less than 45 mg/dL (men); less than 50 mg/dL (women), OR
  * Hypercholesterolemia on stable statin therapy for at least 3 month
* Have a body mass index (BMI) of 18 to 37 kilograms per square meter (kg/m^2), inclusive, at screening

Exclusion Criteria:

* Have known allergies or intolerance to evacetrapib, related compounds
* Have history of recurrent rashes or chronic skin conditions
* Have significant history of or current chronic, active inflammatory conditions
* Have history or current evidence of significant neurological disorder
* Have long-standing diabetes that is insulin requiring
* Have history of or current symptoms of malabsorption syndromes, history of gastric bypass surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Covance Clinical Research Inc, Daytona Beach, Florida
  - Covance, Dallas, Texas
  - Covance Clinical Research Inc, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled into 3 parallel cohorts. Each participant received a single dose, after which PK was evaluated for 7 days, and then continued receiving once daily doses for 12, 24, or 52 weeks. After the last once-daily dose, PK was again evaluated in each participant until the concentration of evacetrapib was too low to be measurable.
Groups:
- Evacetrapib: Multiple Dose 12 Weeks: 130 mg of evacetrapib was administered orally once daily beginning on Day 8 for 12 consecutive weeks.
- Evacetrapib: Multiple Dose 24 Weeks: 130 mg of evacetrapib was administered orally once daily beginning on Day 8 for 24 consecutive weeks.
- Evacetrapib: Multiple Dose 52 Weeks: 130 mg of evacetrapib administered orally once daily beginning on Day 8 for 52 consecutive weeks.
Period: Overall Study
Arm/Group | Evacetrapib: Multiple Dose 12 Weeks | Evacetrapib: Multiple Dose 24 Weeks | Evacetrapib: Multiple Dose 52 Weeks
Started | 30 | 32 | 39
Received at Least 1 Dose of Study Drug | 30 | 32 | 39
Completed | 28 | 29 | 33
Not Completed | 2 | 3 | 6
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Sponsor Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Evacetrapib: Multiple Dose 12 Weeks: 130 mg of evacetrapib administered orally once daily beginning on Day 8 for 12 consecutive weeks
- Evacetrapib: Multiple Dose 24 Weeks: 130 mg of evacetrapib administered orally once daily beginning on Day 8 for 24 consecutive weeks
- Total: Total of all reporting groups
Arm/Group | Evacetrapib: Multiple Dose 12 Weeks | Evacetrapib: Multiple Dose 24 Weeks | Evacetrapib: Multiple Dose 52 Weeks | Total
Number analyzed (Participants) | 30 | 32 | 39 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (14.5) | 51.1 (14.9) | 56.4 (9.4) | 53.8 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 20 | 55
  Male | 13 | 14 | 19 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 6 | 13
  Not Hispanic or Latino | 25 | 30 | 33 | 88
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 8 | 9 | 27
  White | 20 | 23 | 28 | 71
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 32 | 39 | 101

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK) Parameters of Evacetrapib: Area Under the Concentration Versus Time Curve From Time Zero to the Last Time Point With a Measurable Concentration (AUC[0-tlast])
Time Frame: Single-Dose: 1,2,3,4,6,8,12,24,36,48,72,120,168 Hours Postdose; Multiple Dose: Predose, 1,2,3,4,6,8,12,24,36,48,72,120,168 hours; 10,13,17,20,24,29,36,43,50,57, and 71 Days Post Dose
Population: All enrolled participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram∙hour/mililliter (ng∙h/mL)
Groups:
- Evacetrapib: Single Dose, All Participants: A single 130 mg oral dose of evacetrapib was administered on Day 1 to all participants. 130 mg of evacetrapib was administered orally once daily beginning on Day 8 for 12, 24, and 52 consecutive weeks.
Arm/Group | Evacetrapib: Single Dose, All Participants | Evacetrapib: Multiple Dose 12 Weeks | Evacetrapib: Multiple Dose 24 Weeks | Evacetrapib: Multiple Dose 52 Weeks
Number analyzed (Participants) | 101 | 27 | 30 | 29
nanogram∙hour/mililliter (ng∙h/mL) | 14200 (28) | 37400 (43) | 36900 (39) | 44400 (32)

2. Primary Outcome: PK Parameters of Evacetrapib: Maximum Concentration (Cmax)
Time Frame: as for outcome 1
Population: All enrolled participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Evacetrapib: Single Dose, All Participants | Evacetrapib: Multiple Dose 12 Weeks | Evacetrapib: Multiple Dose 24 Weeks | Evacetrapib: Multiple Dose 52 Weeks
Number analyzed (Participants) | 101 | 27 | 30 | 29
nanogram/milliliter (ng/mL) | 1020 (32) | 1690 (41) | 1770 (39) | 1850 (28)

3. Primary Outcome: PK Parameters of Evacetrapib: Terminal Half-life
Time Frame: as for outcome 1
Population: A single terminal half-life estimate was calculated from population PK estimates for apparent clearance and apparent volume of distribution across all participants, based on all available single dose data and multiple dose data.
Measure: Number; unit: Days
Groups:
- Evacetrapib: Single, Multiple Dose 12, 24, and 52 Weeks: A single 130 mg oral dose of evacetrapib was administered on Day 1 to all participants. 130 mg of evacetrapib was administered orally once daily beginning on Day 8 for 12, 24, and 52 consecutive weeks.
Arm/Group | Evacetrapib: Single, Multiple Dose 12, 24, and 52 Weeks
Number analyzed (Participants) | 101
Days | 52.5

4. Secondary Outcome: PD Parameters of Evacetrapib: High Density Lipoprotein Cholesterol (HDL-C) Level
Time Frame: Day -1, Day 8
Population: All enrolled participants in the single dose phase and had evaluable PD data.
Measure: Mean (Standard Deviation); unit: millimole/Liter (mmol/L)
Arm/Group | Evacetrapib: Multiple Dose 12 Weeks | Evacetrapib: Multiple Dose 24 Weeks | Evacetrapib: Multiple Dose 52 Weeks
Number analyzed (Participants) | 30 | 32 | 39
millimole/Liter (mmol/L)
  Single-Dose Phase Day -1 | 1.538 (0.416) | 1.562 (0.395) | 1.670 (0.548)
  Single-dose Phase Day 8 | 1.724 (0.493) | 1.777 (0.443) | 1.772 (0.552)

5. Secondary Outcome: PD Parameters of Evacetrapib: Low-Density Lipoprotein Cholesterol (LDL-C) Level
Time Frame: Day -1, Day 8
Population: All enrolled participants who received at least 1 dose of study drug and had evaluable PD data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Evacetrapib: Multiple Dose 12 Weeks | Evacetrapib: Multiple Dose 24 Weeks | Evacetrapib: Multiple Dose 52 Weeks
Number analyzed (Participants) | 30 | 32 | 39
mmol/L
  Single-Dose Phase Day -1 | 3.711 (0.958) | 3.359 (0.835) | 3.662 (1.039)
  Single-Dose Phase Day 8 | 3.173 (0.872) | 3.152 (0.928) | 3.293 (1.058)

6. Secondary Outcome: PD Parameters of Evacetrapib: Total Cholesterol Level
Time Frame: Day -1, Day 8
Population: All enrolled participants who received at least 1 dose of study drug and had evaluable PD data.
Measure: Mean (Standard Deviation); unit: mmol
Arm/Group | Evacetrapib: Multiple Dose 12 Weeks | Evacetrapib: Multiple Dose 24 Weeks | Evacetrapib: Multiple Dose 52 Weeks
Number analyzed (Participants) | 30 | 32 | 39
mmol
  Single-Dose Phase Day -1 | 5.922 (1.244) | 5.523 (0.736) | 6.015 (1.099)
  Single-Dose Phase Day 8 | 5.577 (1.224) | 5.531 (0.931) | 5.715 (1.179)

7. Secondary Outcome: PD Parameters of Evacetrapib: Triglyceride Level
Time Frame: Day -1, Day 8
Population: All enrolled participants who received at least 1 dose of study drug and had evaluable PD data.
Measure: Mean (Standard Deviation); unit: mmol
Arm/Group | Evacetrapib: Multiple Dose 12 Weeks | Evacetrapib: Multiple Dose 24 Weeks | Evacetrapib: Multiple Dose 52 Weeks
Number analyzed (Participants) | 30 | 32 | 39
mmol
  Single-Dose Phase Day -1 | 1.474 (0.849) | 1.311 (0.815) | 1.485 (0.631)
  Single-Dose Phase Day 8 | 1.482 (1.016) | 1.309 (0.871) | 1.419 (0.681)

ADVERSE EVENTS:
Arm/Group | Evacetrapib: Single Dose, All Participants | Evacetrapib: Multiple Dose 12 Weeks | Evacetrapib: Multiple Dose 24 Weeks | Evacetrapib: Multiple Dose 52 Weeks
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/30 | 0/32 | 5/39
Other Adverse Events (participants affected / at risk) | 12/101 | 13/30 | 17/32 | 22/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evacetrapib: Single Dose, All Participants (N=101) | Evacetrapib: Multiple Dose 12 Weeks (N=30) | Evacetrapib: Multiple Dose 24 Weeks (N=32) | Evacetrapib: Multiple Dose 52 Weeks (N=39)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mycetoma mycotic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evacetrapib: Single Dose, All Participants (N=101) | Evacetrapib: Multiple Dose 12 Weeks (N=30) | Evacetrapib: Multiple Dose 24 Weeks (N=32) | Evacetrapib: Multiple Dose 52 Weeks (N=39)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (4) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (3) | 2 (2) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 4 (5) | 5 (7)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 2 (3)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (4) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 4 (5)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 7 (8) | 4 (6) | 3 (3) | 3 (3)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days